CLINICAL TRIAL: NCT05973123
Title: BLOOM: Boldly Living outdOOrs for Mental Health
Acronym: BLOOM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-38315
Record Dates: First submitted 2023-07-24; First posted 2023-08-02 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Anxiety; Stress Disorder, Posttraumatic; Loneliness; Adverse Childhood Experiences
Keywords: Anxiety; Pediatric Mental Health; Adverse Childhood Experiences
MeSH Terms: conditions — Anxiety Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BLOOM Group Outings (Experimental): 6 weeks of nature based anxiety intervention for families with children who have at least one ACE and higher than average anxiety. Three of the outings will be group outings; the family will conduct 3 of the outings on their own independently.
  Interventions: Behavioral: Group Nature Outings
- BLOOM Independent Outings (Experimental): This group receives text support in going outdoors as a family once a week for 6 weeks to gain skills in managing anxiety.
  Interventions: Behavioral: Family Outings
- Control (No Intervention): Wait listed control. Receives standard of care referral to mental health resources on enrollment. At the end of study receives information on health benefits of being outdoors in nature and an invitation to group outings through the SHINE program at UCSF Benioff Children's Hospital Oakland.

INTERVENTIONS:
Behavioral: Group Nature Outings — A 6 week nature-based intervention for pediatric anxiety. Every other week group outings for families in nature, alternating with every other week nature-based goals for families at home.
  Arms: BLOOM Group Outings
Behavioral: Family Outings — 6 weeks of weekly outings into nature. These will be supported by the research team through a weekly text message and written materials on skill building and activities to do outdoors.
  Arms: BLOOM Independent Outings

SUMMARY:
In 2019, the Office of the California Surgeon General launched the ACEs Aware Initiative in collaboration with the California Department of Health Care Services. This ambitious campaign aims to develop a network of care model of healthcare delivery that explicitly links health resources within communities to clinicians screening patients for ACEs. The ACEs Aware Initiative recognizes nature experiences as one of seven "stress busters." Indeed, California boasts many outdoor resources for clinicians to integrate into the network of care. Through a calming effect on the autonomic nervous system, providing a setting for supportive relationships to develop and physical activity to occur, time in nature may help California prevent, heal and treat ACEs and the clinical sequelae. As one of the most common psychiatric disorders in youth, anxiety remains one of the most important sequelae of ACEs. There is a gap in evidence evaluating nature-based programs for child mental health. This study will evaluate BLOOM [Boldly Living outdOOrs for Mental health], a new intervention which is a modified version of an existing nature-based curriculum called SHINE (Stay Healthy In Nature Everyday) curriculum currently in place at UCSF Benioff Children's Hospital Oakland, which takes youth and their families into nature once a month for stress relief. This new intervention mirrors SHINE except that it will be tailored to children ages 9-12 with a history of ACEs and current anxiety. This study will evaluate the benefits of a group intervention model, an independent nature-outing model, and a comparison to a wait-listed control group. Our goal is to provide a scalable model for low-cost mental health care to the California Department of Health Care Services.

ELIGIBILITY:
Pediatric Inclusion Criteria:

1. Age 9-12 years at enrollment
2. Has an ACE Score of 1 or higher
3. Has a SCARED-P score of 15 or higher
4. Is available to attend three group outings if assigned to group intervention arm.
5. Has a caregiver who is able to consent and attend outings with them.
6. Is able to read, write, and speak English, Spanish or Arabic.
7. Has no serious health conditions that affect their ability to be in nature.
8. Willing to wear a provided electronic sensor continuously for 6 weeks, including sleep, excluding bathing and device recharging time.
9. Have no major changes in their mental health treatment plan during the time of the study.

Caregiver eligibility criteria

1. Able to read, write and speak English, Spanish or Arabic
2. Be at least 18 years old.
3. Have no serious health conditions that affect their ability to be in nature.
4. Is available to attend 6 weekly outings if assigned to group intervention arm.
5. Have a smart phone and be willing to download NatureDose app from NatureQuant.

Exclusion Criteria Child:

1. Concomitant active treatment modification (eg medication changes) for the past month.
2. Unable to attend weekly nature outings if randomized to the group intervention.
3. Physical or health limitation to participating in outdoor activities.
4. Previous SHINE participant.
5. Caregiver unable to consent.
6. Unable to pass short quiz at the end of the assent.
7. Wards of the state who do not have a guardian other than the state who can consent on their behalf.
8. Non-English, Arabic or Spanish speaking participants.
9. Unwilling to use a FitBit.

Exclusion criteria - caregiver

1. Unable to attend weekly nature outings if randomized to the group intervention.
2. Physical or health limitation to participating in outdoor activities.
3. Previous SHINE participant.
4. Unable to provide informed consent.
5. Non-English, Arabic or Spanish speaking participants.
6. Unwilling to use NatureDose app.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 126 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Screen for Child Anxiety Related Emotional Disorders - Parent (SCARED-P) Scores | 6 weeks
  SCARED-P is a measure widely used to assess childhood anxiety. Caregivers will rate pediatric anxiety by taking the SCARED-P assessment, which consists of 41 items that assess a child's recent anxiety symptoms. Participants respond on a 3-point Likert scale of 0 (Not True or Hardly Ever True), 1 (Somewhat or Sometimes True), or 2 (Very True or Often True). Higher scores indicate a higher preponderance of clinically significant anxiety.

SECONDARY OUTCOMES:
Change in Brief Resiliency Screen amongst children | 6 weeks
  Pediatric resilience will be measured, at baseline and at 6 weeks by surveying children directly using the Brief Resiliency Scale. In their systematic review, Windle et al. reviewed 2,979 papers and identified 15 potential scales to measure resiliency in children and adults. Of these, the Brief Resiliency Scale is the only one which had an acceptable Cronbach's alpha (>0.70 and < 0.95 across four different samples), had acceptable criterion validity as it was correlated with Connor-Davidson Resilience Scale and Ego Resiliency Scale. Questions are answered using a five-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Three questions were reverse-scored such that a higher number was associated with greater resilience.

OTHER OUTCOMES:
Change in hair cortisol levels in enrolled children | 6 weeks
  Hair Cortisol levels will be measured at baseline and at 6 weeks for participants who opt into the section of the study. Hair cortisol is a marker of stress over the previous month. Hair cortisol and cortisone levels will be measured by liquid chromatography-tandem mass spectrometry (LC-MS/MS). Samples of hair (5mg, 40-50 stands, 2 cm long) will be obtained from the back of the scalp for consenting child participants.
Change in BMI amongst enrolled children | 6 weeks
  Weight and height measurements will be obtained at baseline and at 6 weeks.
Change in child's nature exposure as measured by GPS coordinates | 6 weeks
  Enrolled children will be asked to wear a FitBit during the course of the study. The FitBit will record the patients GPS coordinates during the course of the 6 weeks of the study. The GPS coordinates will be submitted to the NatureQuant organization without any identifying data. Using satellite and GIS data, NatureQuant will give the research team information about how much vegetation the child was around, and how many parks they visited during the 6 weeks of the study.
Change in caregiver stress as measured by the Perceived Stress Score (PSS-10) | 6 weeks
  Caregivers will fill out the PSS10, a 10-item validated Likert scale, with responses to each item with five options (i.e., never, almost never, sometimes, usually, always). They will fill this out at baseline and at six weeks. A higher score corresponds with higher stress.
Changes in caregiver nature exposure as measured by NatureDose app | 6 weeks
  Enrolled caregivers will be instructed on how to download the NatureDose app on their phones. They will register on the app using a unique research identifier code which does not have personal identifying data on it. The NatureDose app will follow the participant's gps coordinates during the course of the study in order to provide the research team with information about exposure to vegetation and park visits during the six week course fo this clinical trial.

CONTACTS AND LOCATIONS:
Overall Officials: Nooshin Razani, MD MPH, Principal Investigator — UCSF and UCSF Benioff Children's Hospital Oakland
Locations (1):
- UCSF Benioff Children's Hospitals, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No